CLINICAL TRIAL: NCT03896880
Title: Detection of Bloodstream Pathogens in Hematological Malignancies
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Mohammed Tolba, Principle investigator, Assiut University
Other Study IDs: Cancer bloodstream infection
Record Dates: First submitted 2019-03-27; First posted 2019-04-01 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Bloodstream Infection
MeSH Terms: conditions — Sepsis | interventions — Blood Culture; Multiplex Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- blood culture positive: hematological malignancy patients with positive blood culture
  Interventions: Diagnostic Test: blood culture; Other: Anti fungal susceptibility testing or antibiotic susceptibility testing; Other: phenotypic identification methods of the isolated organism by Vitek2 (BioMerieux,France); Other: Identification of the isolated organism by multiplex PCR

INTERVENTIONS:
Diagnostic Test: blood culture — During the febrile episode, two blood samples per patient will draw from two separate sites including central venous catheter if present and directly injected to Bact/Alert® bottles and incubated in Bact/ALERT system instrument (bioMérieux Diagnostics, Lyon, France).
  A-Identification of microorganisms including:
  1. Isolation of microorganisms:
  2. Blood culture samples with positive signals will be cultured on blood agar, chocolate agar , MacConkeys agar and Sabouraud dextrose agar (SDA) plates.
  B-Identification of the bacterial organism
  Pure colonies of isolated microorganisms were identified by:
  Morphology on agar,Gram stain film was made from the growth to identify morphology of the organism ,Biochemical tests
  C-For fungi isolate the following will perform:
  1. Microscopic examination of Lactophenol cotton blue (LCB) wet mounts.
  2. Culture on Brilliance Candida differential agar
Other: Anti fungal susceptibility testing or antibiotic susceptibility testing — isolation of microbes from positive blood culture and anti fungal susceptibility testing or antibiotic susceptibility testing according to isolated microbes by disc diffusion method and Vitek2
  Other Names: antimicrobial susceptibility testing
Other: phenotypic identification methods of the isolated organism by Vitek2 (BioMerieux,France) — The VITEK 2 is an automated microbial identification system that utilizing growth-based technology. With its colorimetric reagent cards, the VITEK 2 offers a state of the art technology platform for phenotypic identification methods.
  Other Names: Vitek2 (BioMerieux,France)
Other: Identification of the isolated organism by multiplex PCR — FilmArray blood culture identification (BCID) is automated multiplex PCR assay, the FilmArray blood culture identification which directly identifies common pathogens, including 7 genera/ species of Gram-positive bacteria, 10 genera/species of Gram-negative bacteria, and 5 species of Candida (as well as 3 resistance determinants) in the positive blood culture bottles. The assay requires about 2 min of hands-on sample processing time and 1 h of instrument time (which includes DNA isolation, amplification, and detection).
  Other Names: FilmArray blood culture identification (BCID); multiplex PCR

SUMMARY:
* To identify the common bacterial and fungal species causing fungemia and bacteremia in hematological malignancies.
* To identify sensitivity pattern for causative microbes.
* Compare culture on ordinary media with Vitek2 (automated microbial identification system) and multiplex polymerase chain reaction (PCR )

DETAILED DESCRIPTION:
Sepsis is a global health problem and an estimated 17 million cases of sepsis occur each year in the world .The early initiation of appropriate antibiotic therapy is determinant for the prognosis and survival of patients with bloodstream infections . Infections in patients suffering from hematological malignancies are a frequent problem, leading to higher mortality and morbidity, increased costs of health care and prolonged duration of hospitalization. Common among these infections are those involving the bloodstream. In febrile neutropenic patients, the attack rate of bloodstream infection was reported to be between 11 and 38% . Hematological malignancies by themselves or by their therapeutic strategies, put patients at risk for infections. Wide use of antibiotics and prophylactic agents in such patients has led to the development of resistance. The general term fungemia describes the presence of a fungal species in the blood while term bacteremia describes the presence of bacterial species in the blood A positive culture may indicate a widespread infection or commonly, the infection of an intravenous catheter .Fungal microbes are abundant in nature and are frequent colonizers on human mucosal surfaces. However, under conditions of impaired immune responses or a break in host barriers, fungi are able to invade normally sterile areas of the human body, where they can cause severe infections that are difficult to recognize and treat and are often ultimately lethal .Indeed, recent epidemiological data show that invasive fungal infections (IFIs) are frequently encountered in clinical practice, with the most common offenders, being Candida spp. and Aspergillus spp. In order to effectively eliminate these infections, early diagnosis and species identification are of paramount importance. Traditional diagnostic methods such as blood culture is still considered the gold standard .Indeed ,novel molecular and non molecular techniques have been developed and currently under clinical evaluation . The VITEK 2 is an automated microbial identification system that utilizing growth-based technology. With its colorimetric reagent cards, the VITEK 2 offers a state of the art technology platform for phenotypic identification methods. The application of the multiplex polymerase chain reaction PCR method in the diagnosis of bloodstream infections is designed to reduce the time for identification of the microorganisms grown from the positive samples to 24-48 hours, as pathogens are identified directly from a positive blood sample

ELIGIBILITY:
Inclusion Criteria:

* hematological malignancy patients on chemotherapy associated with fever

Exclusion Criteria:

* Age below 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hematological malignancy patients with fever
Sampling Method: Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
identify pathogens in positive blood culture in hematological malignancies patients | 1 year
  Examine blood culture to diagnose different species of pathogens including bacteria and fungi responsible for bloodstream infection in hematological malignancies patients.
Antimicrobial susceptibility testing and drug resistance | 1 year
  performance of antimicrobial susceptibility testing (anti fungal susceptibility testing or antibiotic susceptibility testing )of significant bacterial isolates. The goals of testing are to detect possible drug resistance in common pathogens and to assure susceptibility to drugs of choice for particular infections.
prevalence of bloodstream infection in hematological malignancy patients | 1 year
  prevalence of both bacteremia and fungemia in hematological malignancies using blood culture
Time from blood collection to pathogen identification | 1 year
  The hypothesis is that faster identification will lead to faster action.

SECONDARY OUTCOMES:
In-hospital mortality. | 1 year
  Faster treatment is associated with reduced mortality
Rapid diagnosis of bloodstream infections | 1 year
  Compare different methods for rapid identification of blood culture positive results including Vitek2 (BioMerieux,France) and multiplex PCR

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Z Abo krisha, professor, Study Director — Assiut University
Locations (1):
- Assiut university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Salomao R, Diament D, Rigatto O, Gomes B, Silva E, Carvalho NB, Machado FR. Guidelines for the treatment of severe sepsis and septic shock - management of the infectious agent - source control and antimicrobial treatment. Rev Bras Ter Intensiva. 2011 Jun;23(2):145-57. English, Portuguese. PMID 25299714
- [Background] Gedik H, Simsek F, Kanturk A, Yildirmak T, Arica D, Aydin D, Demirel N, Yokus O. Bloodstream infections in patients with hematological malignancies: which is more fatal - cancer or resistant pathogens? Ther Clin Risk Manag. 2014 Sep 17;10:743-52. doi: 10.2147/TCRM.S68450. eCollection 2014. PMID 25258539
- [Background] Yadegarynia D, Tarrand J, Raad I, Rolston K. Current spectrum of bacterial infections in patients with cancer. Clin Infect Dis. 2003 Oct 15;37(8):1144-5. doi: 10.1086/378305. No abstract available. PMID 14523785
- [Background] Brown GD, Denning DW, Gow NA, Levitz SM, Netea MG, White TC. Hidden killers: human fungal infections. Sci Transl Med. 2012 Dec 19;4(165):165rv13. doi: 10.1126/scitranslmed.3004404. PMID 23253612